CLINICAL TRIAL: NCT06355687
Title: The Evaluation of Adding Melatonin to Opioid Free Anesthesia on Postoperative Pain in Obese Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Melatonin in Obese Patients in Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ismail Farid Ibrahim Mahmoud, Assistant Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MD304/2023
Record Dates: First submitted 2024-03-10; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Melatonin group (Active Comparator): Melatonin group: A total of 30 obese patients undergoing laparoscopic cholecystectomy will receive melatonin oral (0.2 mg /kg) 45 minutes before general anesthesia.
  Interventions: Drug: Melatonin
- The Control group (Placebo Comparator): Control group: A total of 30 obese patients undergoing laparoscopic cholecystectomy will receive placebo medication (Vitamin Supplement) 45 minutes before general anesthesia; Control group.
  Interventions: Dietary Supplement: Vitamin Supplement

INTERVENTIONS:
Drug: Melatonin — Obese patients undergoing laparoscopic cholecystectomy will receive melatonin oral (0.2 mg /kg) 45 minutes before general anesthesia.
  Other Names: Circadin
  Arms: The Melatonin group
Dietary Supplement: Vitamin Supplement — Obese patients undergoing laparoscopic cholecystectomy will receive placebo medication (Vitamin Supplement) 45 minutes before general anesthesia.
  Arms: The Control group

SUMMARY:
Opioid free anesthesia (OFA) means a technique in which no intraoperative opioid is administered through any route. Perioperative pain management in an obese patient is challenging. The incidence of respiratory depression is higher in obese patients and is exaggerated with opioids, so the investigators are searching for a drug that has analgesic effect without any effect on respiratory function. In this study, the investigators will add melatonin to OFA in obese patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Obesity leads to a restrictive lung disease, causing reduction in functional residual capacity and total lung compliance.

When an obese patient is supine and anesthetised, the depressant effects of many anesthetic agents and analgesics, particularly opioids, further decrease the lung compliance, leading to increased hypoxemia.

Opioid based general anesthesia in these patients increases the incidence of postoperative respiratory depression, atelectasis, and pneumonia. Also, pain relief with opioids is associated with sedation, hence impeding rapid recovery and early mobilization.

OFA is the use of multimodal or balanced analgesia. The principle of this is to gain additive analgesic effects from different drugs while minimizing side effects, particularly those of opioids. Studies have shown that OFA fast tracks surgery, reduces hospital stay, promotes early mobilization, and enteral nutrition.

Prior studies which investigated opioid free techniques are based on the combination of drugs acting on sympathetic nervous system, perioperative administration of local anesthetics, nonsteroidal anti-inflammatory drugs, and of adjuvant drugs, such as ketamine, magnesium etc.

Laparoscopic surgery is more challenging in obese patients since they have excessive pneumoperitoneal insufflation pressures, longer anesthetic, surgical, and recovery times. Moreover, these procedures are usually done in Trendelenburg position which further leads to increased airway resistance.

Melatonin is mainly secreted from the pineal gland by the suprachiasmatic nucleus. This neurohormone possesses a circadian secretion pattern and regulates the biological clock; it also offers antiemetic, analgesic, and anxiolytic effects. Due to its effect on both acute and chronic pain, melatonin fulfills a beneficial role in reducing postoperative opioid consumption while minimizing nausea and vomiting. In addition, melatonin can be used to moderate the effect of light on the autonomic system.

Several studies have reported that melatonin, as an analgesic, anti-inflammatory, anxiolytic, and anti-agitation premedication, is associated with sedation and anxiolysis without adverse effects on recall and driving performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-45 years.
2. Body Mass Index: Over 30 kg/m2.
3. Physical Status: ASA classification I and II.

Exclusion Criteria:

1. Patient refusal.
2. Age: Less than 18 years, more than 45 years.
3. Patients with known history of allergy towards one of the study drugs.
4. Patients with severe cardiac, respiratory, hepatic or renal disease.
5. Body Mass Index: Under 30 kg/m2.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain. | Will be evaluated postoperatively at time of delivery to Post Anesthesia Care Unit (PACU) (Zero time) and every 5 minutes for 30 minutes.
  Numeric Rating Scale (NRS); is a pain screening tool, commonly used to assess pain severity at that moment in time using a (0-10) scale, with (0) meaning no pain and (10) meaning the worst pain imaginable.

SECONDARY OUTCOMES:
Postoperative Pain. | Will be evaluated at time of 30 minutes after delivery to PACU and hourly for 4 hours.
  Numeric Rating Scale (NRS); is a pain screening tool, commonly used to assess pain severity at that moment in time using a (0-10) scale, with (0) meaning no pain and (10) meaning the worst pain imaginable.
Analgesics usage. | Will be evaluated postoperatively (Zero time) and every 15 minutes for 1 hour.
  The total dose of analgesics consumption was used postoperatively per patient rescue analgesia.
Postoperative nausea and vomiting. | Will be evaluated postoperatively (Zero time) and every 15 minutes for 1 hour.
  The occurrence of postoperative complications including postoperative nausea and vomiting.
Recovery time. | Will be evaluated at time of admission to PACU and every 15 minutes for 1 hour until being discharged from it.
  The time between patient admission to PACU and being discharged from it.
Number of participants with hemodynamic instability. | Will be evaluated at the start of the operation and every 5 minutes throughout the operation until delivery to PACU and every 15 minutes for 1 hour until being discharged from it.
  Intraoperative hemodynamic stability data (Systolic blood pressure; in mmHg, Diastolic blood pressure; in mmHg, and Mean arterial pressure; in mmHg)
Number of participants with hemodynamic instability. | Will be evaluated at the start of the operation and every 5 minutes throughout the operation until delivery to PACU and every 15 minutes for 1 hour until being discharged from it.
  Intraoperative hemodynamic stability data (Heart rate; in beats per second)

CONTACTS AND LOCATIONS:
Overall Officials: Hala GO Salama, MD, Principal Investigator — Faculty of Medicine, Ain Shams University; Reham MU Hashim, MD, Principal Investigator — Faculty of Medicine, Ain Shams University; Walid YO Youssef, MD, Principal Investigator — Faculty of Medicine, Ain Shams University; Diaaeldein MA Haiba, MD, Principal Investigator — Faculty of Medicine, Ain Shams University